CLINICAL TRIAL: NCT00004580
Title: Phase I/II Study of ABT-378/Ritonavir in Protease Inhibitor Experienced HIV-Infected Patients
Brief Title: A Study of ABT-378/Ritonavir Combination in HIV-Infected Patients Who Have Taken Protease Inhibitors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Purpose: Treatment
Other Study IDs: 285B; M97-765
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Nevirapine; HIV Protease Inhibitors; Ritonavir; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Nevirapine

INTERVENTIONS:
Drug: Lopinavir/Ritonavir
Drug: Nevirapine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give ABT-378/ritonavir combination plus nevirapine plus two nucleoside transcriptase inhibitors to HIV-infected patients who previously have taken protease inhibitors. This study also examines how the body handles this combination of anti-HIV drugs.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

- Antiretroviral regimen containing a protease inhibitor and one or two nucleoside reverse transcriptase inhibitors that has not changed in the last 12 weeks.

Patients must have:

- HIV infection with plasma HIV RNA of at least 1,000 copies/ml and less than or equal to 100,000 copies/ml at screening.

Prior Medication:

Allowed:

Naive to or has had less than 8 weeks of at least one nucleoside reverse transcriptase inhibitor and an acceptable regimen of two nucleoside reverse transcriptase inhibitors.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Medications that are contraindicated with ABT-378/ritonavir for the duration of the study, such as midazolam, triazolam, terfenadine, astemizole, cisapride, pimozide, ergotamine and dihydroergotamine.
* Over-the-counter medicine or alcohol, without knowledge or permission of the investigator.

Patients with the following prior conditions are excluded:

* Evidence of acute illness determined by vital signs, physical examination, or laboratory results.
* Clinically significant abnormal ECG results.
* Positive test result for drug abuse with the exception of cannabis, unless the investigator anticipates cannabis use will interfere with compliance with the study.

Prior Medication:

Excluded:

* Investigational drugs with the exception of Amprenavir within 28 days prior to the initiation of study dosing.
* Treatment with a non-nucleoside reverse transcriptase inhibitor.
* Treatment with a protease inhibitor different from the current protease inhibitor for more than 6 weeks prior to current regimen.
* Treatment with more than one protease inhibitor concurrently.

Risk Behavior:

Excluded:

* Active substance abuse, alcohol abuse, psychiatric illness.
* Presumption, by investigator, of poor compliance to regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Pacific Oaks Research, Beverly Hills, California
  - San Francisco Gen Hosp / UCSF AIDS Program, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Rush Presbyterian St Lukes Med Ctr / Sect Infect Dise, Chicago, Illinois
  - Univ North Carolina at Chapel Hill / Dept of Medicine, Chapel Hill, North Carolina
  - Duke Univ Med Ctr / Infectious Disease Clinic, Durham, North Carolina
  - Univ of Cincinnati Med Ctr / Holmes Div Mail Loc 0405, Cincinnati, Ohio
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Infectious Disease Physicians Inc, Annandale, Virginia